CLINICAL TRIAL: NCT04367493
Title: Effects of Chocolate Consumption in the Nutritional State, Quality of Life, Body Composition, Oxidative Stress and Inflammatory Activity in Elderly Patients With Cancer in Palliative Care
Brief Title: Effects of Chocolate Consumption in Elderly Patients With Cancer in Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Nereida Kilza da Costa Lima, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1690/2015
Record Dates: First submitted 2020-04-20; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Nutrition Related Cancer; Aging
Keywords: Palliative Care; Aging
MeSH Terms: interventions — Chocolate

STUDY DESIGN:
Intervention Model Description: Comparative, randomized, non-blind intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Group 55% cocoa intervention (Experimental): 55% cocoa intervention
  Interventions: Dietary Supplement: Chocolate
- 2. Group White Chocolate (Experimental): White chocolate
  Interventions: Dietary Supplement: Chocolate
- 3. Control Group (No Intervention): Control Group

INTERVENTIONS:
Dietary Supplement: Chocolate — 25 g of chocolate by day for 4 weeks
  Arms: 1. Group 55% cocoa intervention; 2. Group White Chocolate

SUMMARY:
Elderly patients with advanced cancer stage constitute an important demand for palliative care, a scenario in which metabolic and nutritional status changes may be present.

The aim of this study was to evaluate the effects of chocolate consumption for 4 continuous weeks on nutritional status, quality of life, body composition, oxidative stress and inflammatory activity of elderly cancer patients in palliative care.

DETAILED DESCRIPTION:
Clinical trial designed as a comparative, randomized, non-blind intervention study involving elderly patients with cancer and palliative care in outpatient follow-up at the University Hospital of the Ribeirão Preto Medical School - University of São Paulo. Patients were randomized into 3 blocks of 15 subjects in the control (CG), 55% cocoa intervention (GI1) and white chocolate (GI2) intervention groups. The volunteers were evaluated before and after 4 weeks (28 days) for clinical and laboratory nutritional parameters, quality of life analysis and presence and grading of symptoms. The nutritional status of the patients was evaluated using the Mini Nutritional Assessment (MNA) and the current and usual food intake through the 24-hour recall survey (IR24h) and the food frequency questionnaire (FFQ), respectively. The body mass index (BMI), arm circumference and calf circumference of the volunteers were obtained and the body composition was evaluated by the deuterium oxide method. The inflammatory profile was analyzed by serum interleukin 6 levels and the antioxidant capacity was evaluated by the quantification of reduced glutathione (GSH) and ascorbic acid. Serum lipid peroxidation was measured by determining malonaldehyde levels and the presence and quantification of damage to genetic material by 8-hydroxy-2'-deoxyguanosine levels. To analyze quality of life, the European Organization for Cancer Research and Treatment (EORTC) - Quality of Life Questionnaire (QLQ) - C30 was administered and the Edmonton Symptom Assessment System (ESAS) scale was used to assess the frequency and intensity of symptoms. Data were analyzed by SAS Statistical Software (version 9.3; SAS Institute, Inc. Cary, NC) and R Core Team (2016). Initially, a descriptive analysis of the data was performed. Chi-square test was used to evaluate categorical variables. For the comparison between the groups at each moment and between the moments in each group was used linear regression model with mixed effects. The significance level established was <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients with cancer and palliative care in outpatient follow-up, with Karnofsky Palliative Scale (KPS) of 60% or more

Exclusion Criteria:

* Karnofsky Palliative Scale (KPS) of less than 60%

Ages: 60 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Nutritional Status | 4 weeks
  Evaluation by Mini Nutritional Assessment, by the 24-hour Recall Survey, and by the Food Frequency Questionnaire at the basal moment and after 4 weeks of intervention.
Change in Food Ingestion | 4 weeks
  Evaluation of ingestion by the 24-hour Recall Survey and by the Food Frequency Questionnaire at the basal moment and after 4 weeks of intervention.
Change in Body Composition | 4 weeks
  Body composition was evaluated by the deuterium oxide method at the basal moment and after 4 weeks.
Change in Level of Quality of Life | 4 weeks
  The European Organization for Cancer Research and Treatment Questionnaire was administered before and after the intervention of 4 weeks.

SECONDARY OUTCOMES:
Change in the measurements of oxidative stress | 4 weeks
  The antioxidant capacity was evaluated by the quantification of reduced glutathione and ascorbic acid. Serum lipid peroxidation was measured by determining malonaldehyde levels and the presence and quantification of damage to genetic material by 8-hydroxy-2'-deoxyguanosine levels. All measurements were performed before and after 4 weeks of intervention.
Change in inflammatory status | 4 weeks
  Inflammatory status was evaluated by serum Interleukin 6 levels and C Reactive Protein evaluated before and after the intervention.

REFERENCES:
- [Derived] Vettori JC, da-Silva LG, Pfrimer K, Jordao AA, Louzada-Junior P, Moriguti JC, Ferriolli E, Lima NKC. Effect of chocolate on older patients with cancer in palliative care: a randomised controlled study. BMC Palliat Care. 2022 Jan 4;21(1):5. doi: 10.1186/s12904-021-00893-1. PMID 34980096